CLINICAL TRIAL: NCT04423692
Title: Knowledge About Covid-19 Infection in Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Researcher at national research center, egypt, Aljazeera Hospital
Other Study IDs: Knowledge about covid 19
Record Dates: First submitted 2020-06-07; First posted 2020-06-09 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Viral Infection
MeSH Terms: conditions — Virus Diseases | interventions — Counseling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women with abnormal labs: Mothers who have abnormal labs during pregnancy with abnormal coagulation profile
  Interventions: Other: labs

INTERVENTIONS:
Other: labs — A group of questions to women regarding Corona with laboratory finding suggestive of covid 19 and coagulopathy
  Other Names: Questions and counseling

SUMMARY:
Covid 19 is a pandemic infection developed in late 2019

DETAILED DESCRIPTION:
It developed in China Then spread worl wide

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

* non pregnant women

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant 6and women who have children
Study Population: Pregnant women at any GA
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
The number of pregnant women who have knowledge about covid-19 | one month
  The proper knowledge about covid-19

CONTACTS AND LOCATIONS:
Locations (1):
- Aljazeera( Al Gazeera) hospital, Giza, Egypt